CLINICAL TRIAL: NCT05479474
Title: Platelet Rich Plasma Testis
Brief Title: Platelet Rich Plasma Testis Treatment for Infertile Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Eisenberg, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65917
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Male Infertility; Nonobstructive Azoospermia; Azoospermia
MeSH Terms: conditions — Infertility, Male; Azoospermia, Nonobstructive; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet rich plasma treatment arm (Experimental): After consent in obtained, the patient will undergo a blood draw (12 tsp) to prepare the PRP infusion. The use of a centrifuge and an Arteriocyte Magellan kit are necessary for the PRP preparation. After injection of local anesthesia, PRP will be injected into each testicle.
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: Platelet rich plasma — Patients will undergo a blood draw (12 tsp) to prepare the PRP infusion. The use of a centrifuge and an Arteriocyte Magellan kit are necessary for the PRP preparation. After injection of local anesthesia, PRP will be injected into each testicle.
  * On the third month after the testicular PRP procedure, a TESE will be performed
  * If the procedure is successful a new IVF cycle using the sperm procured from the procedure will be done.

SUMMARY:
Investigate the effect of intratesticular injection of autologous platelet rich plasma (PRP) on sperm retrieval rates and IVF outcomes in infertile men who already underwent a negative sperm retrieval. Currently, there is no alternative treatment after failed TESE. Prior series suggest that intratesticular PRP injections may improve TESE outcomes. We hope to determine whether PRP is an effective treatment for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 18 diagnosed with NOA and at least one failed TESE, negative mapping or negative biopsy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
sperm present | 3 months after PRP injection
  A TESE procedure will be performed to determine if sperm are present

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Urology Clinic, Stanford, California, United States